CLINICAL TRIAL: NCT01111955
Title: A Double-blind, Placebo-Controlled, Parallel-group, Randomized, Multiple-Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamic Effects of BMS-823778 in Subjects With Type 2 Diabetes Who Have Inadequate Glycemic Control on Either Diet and Exercise Alone or on a Background of Metformin
Brief Title: Safety Study of BMS-823778 in Subjects With Type 2 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MB121-002
Record Dates: First submitted 2010-04-26; First posted 2010-04-28 (Estimated); Last update posted 2015-10-12 (Estimated); Status verified 2015-09

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — BMS-823778; Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- BMS-823778 (2 mg) (Active Comparator): + metformin
  Interventions: Drug: BMS-823778; Drug: Metformin
- BMS-823778 (10 mg) (Active Comparator): + metformin
  Interventions: Drug: BMS-823778; Drug: Metformin
- BMS-823778 (20 mg) (Active Comparator): + metformin
  Interventions: Drug: BMS-823778; Drug: Metformin
- Placebo (Placebo Comparator): + metformin
  Interventions: Drug: Placebo; Drug: Metformin

INTERVENTIONS:
Drug: BMS-823778 — Capsules, Oral, 2 mg, once daily, 28 days
  Arms: BMS-823778 (2 mg)
Drug: BMS-823778 — Capsules, Oral, 10 mg, once daily, 28 days
  Arms: BMS-823778 (10 mg)
Drug: BMS-823778 — Capsules, Oral, 20 mg, once daily, 28 days
  Arms: BMS-823778 (20 mg)
Drug: Placebo — Capsules, Oral, 0 mg, once daily, 28 days
  Arms: Placebo
Drug: Metformin — Capsules, Oral, ≥ 1500 mg, once daily, 28 days

SUMMARY:
The purpose of this study is to assess the safety, tolerability and pharmacodynamic effects on fasting plasma glucose (FPG).

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus
* Drug naive or on stable metformin therapy
* HbA1c 7-10%
* FPG ≤ 240mg/dL

Exclusion Criteria:

* History of myocardial infarction, coronary angioplasty or bypass grafts, valvular disease or repair, unstable angina pectoris, transient ischemic attack, or cerebrovascular accidents within six months prior to entry into the study
* Congestive heart failure
* Active liver disease
* Impaired renal function
* Hepatitis C, B and HIV

This list is not inclusive; additional information is provided in the protocol

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2010-07; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Lowering of fasting plasma glucose (FPG) throughout the study to see if there is a decrease from baseline | Within 28 days following dosing

SECONDARY OUTCOMES:
Pharmacokinetics (measuring trough concentrations) | On days 7, 14 and 28
Pharmacodynamics (measuring daily glucose, glucose AUC, HbA1c, lipid profiles, HPA markers, free testosterone, and SHBG) | Within 28 days following dosing

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (14):
- United States (3):
  - Farid Marquez, Md, Hialeah, Florida
  - Capital Clinical Reserch Center, Olympia, Washington
  - Aurora Advanced Healthcare, Milwaukee, Wisconsin
- Australia (3):
  - Local Institution, Blacktown, New South Wales
  - Local Institution, Box Hill, Victoria
  - Local Institution, Freemantle, Western Australia
- Canada (8):
  - Local Institution, Surrey, British Columbia
  - Local Institution, Winnipeg, Manitoba
  - Local Institution, Bathurst, New Brunswick
  - Local Institution, St. John's, Newfoundland and Labrador
  - Local Institution, Thornhill, Ontario
  - Local Institution, Mirabel, Quebec
  - Local Institution, Québec, Quebec
  - Local Institution, Saskatoon, Saskatchewan

REFERENCES:
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx